CLINICAL TRIAL: NCT04939714
Title: Mastering the Challenges of Dementia Family Caregiving in a Time of COVID-19: An Online Course
Brief Title: Caregiving During Crisis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Carolyn Clevenger, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001424; 3P30AG064200-02S1 (NIH)
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Caregiver Stress Syndrome
Keywords: Dementia family caregiver; Online education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducational Intervention (Experimental): Caregivers receiving the psychoeducational intervention immediately.
  Interventions: Behavioral: Psychoeducational Intervention
- Waitlist (No Intervention): Caregivers on a waitlist to receive the psychoeducational intervention after a waiting period of 8 weeks.

INTERVENTIONS:
Behavioral: Psychoeducational Intervention — The intervention is an online course providing education and training to caregivers over an 8 week period. The self-paced course provides information on caregiving for a PLWD during a pandemic, navigating the health care system for a PLWD, and managing daily life (including self-care).
  Arms: Psychoeducational Intervention

SUMMARY:
This study will test a prototype pandemic caregiver training and education course designed for caregivers of persons living with dementia (PLWD). Participants will be randomized to take the course immediately or to take the course after completion of an 8-week waiting period.

DETAILED DESCRIPTION:
Family caregivers, the backbone of care for the upwards of 7 million community-dwelling individuals living with Alzheimer's disease in the U.S., provide at least 85% of the care these individuals receive, at some risk to their own well-being, and are instrumental in navigating healthcare systems. Without their care, it is almost certain that persons living with dementia (PLWD) would have much higher rates of acute and emergency care use than their age-matched peers, perilous venues for them in the best of times, potentially deadly during this pandemic. With coronavirus disease 2019 (COVID-19) restrictions, the amount of care they provide and the expertise needed to provide the care will increase. Typically, caregivers are strangers in healthcare and pandemic landscapes, but they are now called on to enact home care and safety measures and navigate an intricate, complex, and opaque system without the benefit of a compass or a translator, and largely without understanding their role in or having the skills for navigating the system. A variety of interventions have demonstrated benefit in enhancing caregivers' caregiving capacities, with resulting positive outcomes for both caregivers and care recipients. Only a few of these useful interventions, Tele-Savvy among them, have employed distance delivery means, thus enabling rural caregivers and others precluded by circumstance from attending in-person programs to take part in the intervention programs.

The study will assess a psychoeducational intervention for dementia caregivers. Participating caregivers will be randomized to immediately enroll in the study intervention or to be in a waitlist group that will begin the intervention 8 weeks later. Participants will complete interviews at baseline and after the 8-week study period.

ELIGIBILITY:
Inclusion Criteria:

* Providing care for a family member or friend with a confirmed diagnosis of dementia
* Lives in the community
* Co-resides with the PLWD
* Is the main caregiver for the PLWD
* Has access to a computer with internet service
* Can read and understand English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Clevenger, DNP, APRN, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be made available for sharing, after deidentification.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be available for sharing beginning 3 months and ending 5 years following article publication.
Access Criteria: Individual participant data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve aims in the approved proposal. Proposals should be directed to carolyn.clevenger@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website.

RESULTS

PARTICIPANT FLOW:
Groups:
- Psychoeducational Intervention Immediately: Caregivers receiving the psychoeducational intervention immediately.
- Psychoeducational Intervention After Waiting Period: Caregivers receiving the psychoeducational intervention after a waiting period of 8 weeks.
Period: Overall Study
Arm/Group | Psychoeducational Intervention Immediately | Psychoeducational Intervention After Waiting Period
Started | 50 | 50
Completed Week 8 Assessment | 38 | 38
Completed (Completed Week 16 Assessment) | 33 | 30
Not Completed | 17 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychoeducational Intervention Immediately | Psychoeducational Intervention After Waiting Period | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age is missing for one caregiver
  years
    number analyzed (Participants) | 49 | 50 | 99
    (all) | 65.245 (8.971) | 63.800 (11.772) | 64.515 (10.451)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 42 | 40 | 82
  Male | 6 | 10 | 16
  Missing response | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 48 | 45 | 93
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 40 | 80
  African American/Black | 8 | 7 | 15
  Asian | 1 | 1 | 2
  Other | 0 | 1 | 1
  Missing response/did not wish to answer | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100
Highest Education Level [Count of Participants; unit: Participants]
  High school/General Educational Development (GED) certificate | 1 | 0 | 1
  Some college | 13 | 8 | 21
  College graduate | 14 | 16 | 30
  Graduate degree | 21 | 26 | 47
  Missing response | 1 | 0 | 1
Employed Outside of the Home [Count of Participants; unit: Participants]
  No | 33 | 35 | 68
  Yes | 16 | 15 | 31
  Missing response | 1 | 0 | 1
Sexual Orientation [Count of Participants; unit: Participants]
  Bisexual | 0 | 1 | 1
  Gay | 0 | 0 | 0
  Lesbian | 1 | 0 | 1
  Heterosexual | 22 | 23 | 45
  Missing response | 27 | 26 | 53
Geographic Area of Residence [Count of Participants; unit: Participants]
  Urban | 17 | 15 | 32
  Suburban | 22 | 30 | 52
  Rural | 10 | 5 | 15
  Missing response | 1 | 0 | 1
Care Provided for Spouse [Count of Participants; unit: Participants]
  No | 25 | 27 | 52
  Yes | 25 | 23 | 48
Age of Person Cared For [Mean (Standard Deviation); unit: years] — Population: Age is missing for one person receiving care
  years
    number analyzed (Participants) | 49 | 50 | 99
    (all) | 77.939 (9.286) | 78.560 (7.077) | 78.253 (8.208)
Reside in Same House as Person Receiving Care [Count of Participants; unit: Participants]
  No | 9 | 12 | 21
  Yes | 40 | 38 | 78
  Missing response | 1 | 0 | 1
Person Cared for Diagnosed with Dementia [Count of Participants; unit: Participants]
  No | 5 | 3 | 8
  Yes | 44 | 47 | 91
  Missing response | 1 | 0 | 1
Stage of Dementia of Person Cared For [Count of Participants; unit: Participants]
  Early Stage - A person may function independently but is having memory lapses | 5 | 5 | 10
  Middle Stage - greater difficulty performing tasks but still remembers significant life details | 32 | 33 | 65
  Late Stage - loses ability to respond with environment/needs extensive help with daily activities | 7 | 9 | 16
  No known diagnosis of dementia | 6 | 3 | 9
Amount of Help From Friends and Family [Count of Participants; unit: Participants]
  A great deal of help | 8 | 11 | 19
  Some help | 9 | 10 | 19
  A little help | 6 | 10 | 16
  Not much help | 2 | 2 | 4
  Almost no help | 0 | 1 | 1
  Missing response | 25 | 16 | 41
Amount of Strife [Count of Participants; unit: Participants] — Participants were asked "Thinking about your family and friends and about your caregiving and support responsibilities, how much strife and disagreement have family and friends added to the difficulties you may face in your overall caregiving experience?"
  Participants
    They have only been helpful | 16 | 12 | 28
    Hardly any problems | 16 | 21 | 37
    Occasional Strife | 11 | 11 | 22
    Some serious difficulties | 6 | 2 | 8
    A main source of difficulties | 0 | 4 | 4
    Missing response | 1 | 0 | 1
Also Provide Care to Others [Count of Participants; unit: Participants] — Participants were asked "Are there others in your family or among your friends and neighbors for whom you also feel responsible to provide care or other kinds of support (e.g. financial, legal, emotional, logistical, etc.)?"
  Participants
    No | 25 | 28 | 53
    Yes | 24 | 22 | 46
    Missing response | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiologic Studies - Depression (CES-D) Scale Score
Description: The CES-D is a 20-item self-report instrument asking respondents if they have experienced symptoms of depression during the past week. Responses are given on a scale of 0 to 3 where rarely is scored as 0 and most of the time is scored as 3. Total scores range from 0 to 60 and higher scores indicate greater symptoms of depression.
Time Frame: Baseline, Week 8
Population: This analysis includes participants who attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Waitlist Control Group: Caregivers on a waitlist to receive the psychoeducational intervention after a waiting period of 8 weeks.
Arm/Group | Psychoeducational Intervention | Waitlist Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline | 11.7 (8.8) | 11.8 (8.0)
  Week 8: number analyzed (Participants) | 38 | 38
  Week 8 | 10.4 (8.7) | 14.6 (9.6)

2. Primary Outcome: State-Trait Anxiety Inventory (STAI) Score
Description: The STAI is a 20-item self-report scale of positive and negative anxiety experiences. Responses are given on a 4-point scale where 1 = not at all and 4 = very much so. Total scores range from 20 to 80 and higher scores indicate greater anxiety.
Time Frame: Baseline, Week 8
Population: This analysis includes participants who attended the indicated study visits and who provided complete information for the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychoeducational Intervention | Waitlist Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline | 29.7 (8.5) | 33.7 (9.1)
  Week 8: number analyzed (Participants) | 36 | 38
  Week 8 | 32.6 (10.4) | 38.2 (12.5)

3. Primary Outcome: Perceived Stress Scale (PSS-14) Score
Description: The Perceived Stress Scale includes 14 items assessing self-reported caregiving stress. Responses are given on a 5-point scale where 0 = never and 4 = very often. Total scores range from 0 to 56 and higher values indicate greater perceived stress.
Time Frame: Baseline, Week 8
Population: This analysis includes participants who attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychoeducational Intervention | Waitlist Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline | 22.3 (7.9) | 22.4 (7.3)
  Week 8: number analyzed (Participants) | 38 | 38
  Week 8 | 21.7 (7.1) | 23.1 (8.1)

4. Primary Outcome: Revised Memory and Behavior Problem Checklist (RMBPC) Frequency Score
Description: The RMBPC is a 24-item scale reporting on frequency of disturbing care recipient behaviors and severity or caregiver reactions to these behaviors. Respondents indicate how frequently problems have occurred on a 5-point scale where 0 = never occurred and 4 = daily or more often. Total frequency scores range from 0 to 96 with higher scores indicating greater frequency of memory and behavior problems exhibited by the person living with dementia (PLWD).
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychoeducational Intervention | Waitlist Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline | 39.3 (11.0) | 40.1 (12.4)
  Week 8: number analyzed (Participants) | 38 | 37
  Week 8 | 39.0 (11.8) | 38.2 (13.4)

5. Primary Outcome: Revised Memory and Behavior Problem Checklist (RMBPC) Reaction Score
Description: The RMBPC is a 24-item scale reporting on frequency of disturbing care recipient behaviors and severity or caregiver reactions to these behaviors. Respondents indicate the degree to which problems have bothered or upset them on a 5-point scale where 0 = not at all and 4 = extremely. Total reaction scores range from 0 to 96 with higher scores indicating more bothered or upset by memory and behavior problems exhibited by the PLWD.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychoeducational Intervention | Waitlist Control Group
Number analyzed (Participants) | 49 | 50
score on a scale
  Baseline | 15.3 (8.9) | 16.3 (11.7)
  Week 8: number analyzed (Participants) | 38 | 36
  Week 8 | 14.9 (9.0) | 16.3 (14.1)

6. Primary Outcome: Zarit Burden Interview Score
Description: The Zarit Burden Interview is a 22-item scale of objective and subjective caregiver burden. Responses are given on a 5-point scale where 0 = never and 4 = nearly always. Total scores range from 0 to 88 where higher scores indicate greater feelings of being burdened with providing care.
Time Frame: Baseline, Week 8
Population: This analysis includes participants who attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychoeducational Intervention | Waitlist Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline | 33.9 (12.6) | 37.9 (14.1)
  Week 8: number analyzed (Participants) | 38 | 38
  Week 8 | 33.1 (13.1) | 39.0 (13.2)

7. Primary Outcome: Caregiver Mastery Scales - Competency Score
Description: The Caregiving Mastery instrument assesses caregiver mastery of 3 different realms of caregiving situations: Relational Deprivation, Caregiving Competence, and Management of Situation. The Caregiving Competence section includes 4 items are responded to on a 4-point scale where 1 = not at all and 4 = completely. Total scores range from 4 to 16 where higher scores indicate greater feelings of mastery of caregiving.
Time Frame: Baseline, Week 8
Population: This analysis includes participants who attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychoeducational Intervention | Waitlist Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline | 12.9 (1.8) | 12.5 (1.9)
  Week 8: number analyzed (Participants) | 38 | 38
  Week 8 | 13.4 (1.6) | 12.6 (1.7)

8. Primary Outcome: Caregiver Assessment of Behavioral Skill - Self-report Score
Description: The Caregiver Assessment of Behavioral Skill - Self-report instrument is a 17-item caregiver self-assessment of perceived capacity to manage care situations. Responses are given on a 3-point scale where 0 = seldom true and 3 = true most of the time, for behaviors exhibited by or relevant to the PLWD. Total scores range from 0 to 51 where higher scores indicate perceived ability to manage providing care.
Time Frame: Baseline, Week 8
Population: This analysis includes participants who attended the indicated study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychoeducational Intervention | Waitlist Control Group
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline | 14.3 (5.9) | 15.1 (5.7)
  Week 8: number analyzed (Participants) | 38 | 38
  Week 8 | 14.1 (6.7) | 14.4 (4.9)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Week 16.
Arm/Group | Psychoeducational Intervention Immediately | Psychoeducational Intervention After Waiting Period
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT04939714/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04939714/ICF_001.pdf